CLINICAL TRIAL: NCT02902393
Title: Interest of Thromboelastography (ROTEM) as a Biomarker of Revascularisation in Stroke
Acronym: ROTEMPredict
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 15-202
Record Dates: First submitted 2016-09-07; First posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Stroke
Keywords: Fibrinolysis; tPA
MeSH Terms: conditions — Stroke | interventions — Thrombelastography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Success of revascularisation
  Interventions: Biological: Thromboelastography

INTERVENTIONS:
Biological: Thromboelastography

SUMMARY:
Revascularisation using recombinant tPA is the reference treatment of stroke. However, the efficacy of fibrinolysis is about 50%. Several factors, including the size of thrombus, have been associated with revascularisation efficacy.

The aim of this prospective study is to evaluate ex vivo the effect of tPA in patients with stroke with thromboelastography and to correlate results with the clinical outcome of patients. Results may predict revascularisation in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patient (> 18 years) with a neurological deficit compatible with a neurovascular pathology eligible for fibrinolysis rtPA and having a proximal occlusion of the middle cerebral artery (segment M1 / M2) or basilar trunk objectified brain imaging (MRI angiography or angio CT).

Exclusion Criteria:

* Any patient with major comorbidity, a pathology of hemostasis or anticoagulant treatment (vitamin K antagonist (VKA), direct oral anticoagulant).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients meeting the eligibility criteria will be invited to participate in the study . Patients will be recruited to emergencies CHU Caen and Saint Joseph Hospital. The goal is to recruit patients with neurological defect consistent with a neurovascular pathology eligible for thrombolysis with tPA.
  With the admission of patients, blood samples are routinely made . For this study, the investigators will add one citrated 5 mL tube. An information letter and consent form will be given to the patient.
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-06 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of revascularisation 24 hours after tPA injection using CT scan or MRI | 24 hours

SECONDARY OUTCOMES:
Clinical evaluation using NIHSS scale | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Richard MACREZ, PhD, Principal Investigator — University Hospital, Caen
Locations (1):
- University Hospital, Caen, Calvados, France